CLINICAL TRIAL: NCT03683121
Title: Effect of Different Follow-up Methods on Compliance and Prognosis of NSBB Secondary Prevention of Cirrhosis With Gastroesophageal Varices Bleeding
Brief Title: The Compliance and Prognosis of NSBB Secondary Prevention of Cirrhosis With Gastroesophageal Varices Bleeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, ChenMingkai, Chief physician of Department of Gastroenterology I, Renmin Hospital of Wuhan University
Other Study IDs: ChenMingkai
Record Dates: First submitted 2018-09-15; First posted 2018-09-25 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Esophageal Varices Bleeding
Keywords: Esophagogastric variceal hemorrhage; cirrhosis; secondary prevention; Non-selective beta blocker; compliance
MeSH Terms: conditions — Fibrosis; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- the traditional follow-up group: The dose and notes for the use of the Non-selective beta blockers were informed during outpatient follow-ups for the patients with a history of esophageal variceal bleeding
- Non-traditional follow-up: The dose and notes for the use of the Non-selective beta blockers were informed during telephone or WeChat follow-ups for the patients with a history of esophageal variceal bleeding
- Combine of Group1 and Group2: The dose and notes for the use of the Non-selective beta blockers were informed during outpatient follow-ups for the patients with a history of esophageal variceal bleeding,and the patients were followed up by telephone or WeChat again on the same day.

SUMMARY:
Non-selective beta blockers are commonly used drugs for primary prevention and secondary prevention in patients with cirrhotic decompensated esophageal varices bleeding，the basic heart rate, blood pressure and condition of different patients have individual differences.This paper mainly discusses the compliance of patients taking NSBB under different follow-up methods and analyze the factors affecting patient compliance.

DETAILED DESCRIPTION:
Esophagogastric variceal hemorrhage is a common complication of decompensated liver cirrhosis and the rate of rebleeding after hemostasis is high.Effective secondary prevention reduces the risk of rebleeding.Non-selective beta blockers are commonly used drugs for secondary prevention.Clinically, there is a great difference in the compliance of patients taking non-selective beta receptor blockers.In this study, the enrolled patients were divided into three groups: the traditional follow-up group (face-to-face interview);Non-traditional follow-up (WeChat, telephone, etc.);Traditional and non-traditional methods of follow-up were combined in the group.The investigators collected the basic data before the patients were enrolled, adjusted the medication dosage according to the patients' condition during the follow-up period, and recorded the treatment during the follow-up period, and analyzed the factors influencing the patients' compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. All cases met the diagnostic criteria for cirrhosis
3. All patients were confirmed to be combined with esophageal and gastric varices through endoscopy or portal vein CTA or abdominal CT, and had at least one history of esophageal and gastric varices rupture and bleeding. Child-pugh was graded as A/B.
4. All patients had basal heart rate greater than 60 beats/min and systolic pressure greater than 90mmhg.

Exclusion Criteria:

1. Patients with liver cancer or other gastrointestinal tumors
2. Patients with splenomegaly due to extrahepatic portal hypertension and noncirrhosis
3. Patients with basal heart rate less than 55 beats/min or systolic pressure less than 90mmhg
4. There are patients with NSBB contraindications such as severe cardiac insufficiency, cardiogenic shock, sinus bradycardia and morbid sinus syndrome, severe ventricular conduction block, bronchial asthma, etc.
5. Patients with other diseases other than liver cirrhosis should take beta blockers (such as coronary heart disease, arrhythmia, etc.).
6. Patient data is incomplete, data cannot be collected and counted
7. Patients who do not agree with secondary prevention after informing them about the adverse reactions associated with medication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient was diagnosed with liver cirrhosis in the investigator's hospital or the outer court and had a history of esophageal variceal rupture and bleeding before into the group
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate compliance ratio after treatment with NSBBs | 10 months
  In this single-center study, 83 patients were included, including 9 cases lost to follow-up, 1 case died, and 1 case was excluded from liver cancer. a total of 72 cases were included, with an average follow-up time of 185.3 days.Among the 72 patients who were not lost to follow-up, 40 NSBBs patients had good medication compliance, and 34 patients achieved heart rate response (34/40,85.0%).

SECONDARY OUTCOMES:
Different follow-up methods were used to guide non-hospitalized patients to take medication in NSBBs, and the compliance of patients with NSBBs and its influencing factors were analyzed | 10 months
  Three follow-up methods guided secondary prevention of NSBBs, and the compliance of patients in the remote platform follow-up group and the outpatient clinic combined with the remote platform follow-up group was higher than that in the outpatient follow-up group (P < 0.05).There was no statistically significant difference in patient compliance between the remote platform follow-up group and the outpatient combined remote platform follow-up group.In outpatient follow-up, there was a statistically significant difference between the subgroup of NSBBs with good compliance and poor compliance, and the local resident patients had better compliance
The compliance of gastroscopy and bleeding of esophageal and gastric varices during the follow-up period were analyzed | 10 months
  The compliance of the subgroup of NSBBs with good medication compliance was 30/40 (75.0%) during the follow-up period of gastroscopy, and 14/30 (46.7%) after gastroscopy was followed up for sequential endoscopic treatment.Poor compliance of NSBBs subgroup during the follow-up period, the compliance of gastroscopy was 7/32 (21.9%), and 3/7 (42.9%) after gastroscopy, sequential treatment under endoscopy.During the follow-up period, the subgroup with good medication compliance of NSBBs had higher compliance with gastroscopy than the subgroup with poor medication compliance (P=0.000).

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided